CLINICAL TRIAL: NCT03916874
Title: A Longitudinal Study to Understand How Gut Microbes Contribute to Maintaining Health During Pregnancy and Early Life.
Brief Title: The Pregnancy & Early Life Study
Acronym: PEARL
Status: Active, not recruiting | Type: Observational
Sponsor: Quadram Institute Bioscience (Other)
Collaborators: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: QIB02/2018
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — faeces, urine, skin swabs, vaginal swabs, breast milk (optional), blood (optional)
Oversight: Data Monitoring Committee: Yes | US Export: No

GROUPS / COHORTS (1):
- Pregnant females and her newborn.: A longitudinal study of one cohort of 250 pregnant females less than 22 weeks gestation and her newborn. Swabs and samples (low vaginal, skin, urine, blood and stool) will be requested at one time point during each trimester from the participant. In addition, there are three different questionnaires at trimester 2.

SUMMARY:
The gut is home to a diverse and dynamic microbial community, termed the microbiota. The microbiota is essential for health and wellbeing and is involved in acquisition of nutrients and energy from the diet, optimisation of the immune system, and resistance against invading pathogens. Critically, in both new mothers and their babies, any disturbance of the microbiota (caused, for example, by antibiotics, delivery mode [vaginal/Caesarean section], or dietary change), has the potential to increase the risk that the baby might subsequently develop allergic-type disorders, infections, and chronic intestinal diseases.

Early life is a key period of development, but the investigators need a clearer understanding of how maternal factors and transmission of beneficial microbes from mother to baby influence the development of a healthy infant microbiota. This is only possible through longitudinal studies, where the profiles of microbiota from cohorts of mothers and their babies are correlated with routine and more specific clinical data (i.e. antibiotics and diet) throughout pregnancy and into early life.

In order to achieve the aims of the study, the Quadram Institute Bioscience (QIB) will work in collaboration with the Norfolk & Norwich University Hospital (NNUH) to recruit 250 pregnant female participants. Study duration will be approximately 31 months and during this time, the investigators will ask the participants to collect urine and stool samples and low vaginal and skin swabs. Blood samples and breast milk are optional. From her newborn, investigators will ask the participant to collect a meconium and stool samples and skin swabs. The participant will complete three different types of questionnaires for herself and her newborn over 31 months. This study is fully funded by the Biotechnology and Biological Sciences Research Council (BBSRC).

DETAILED DESCRIPTION:
The gut is home to a diverse and dynamic microbial ecosystem, termed the microbiota. These microbes provide their host with various beneficial effects including acquisition of additional nutrients and energy from dietary components, optimal development of the immune system, and resistance against invading pathogenic microbes, and are thus critical for health. As the neonatal gut is essentially sterile at the outset, these beneficial microbes and their associated functions are acquired after initial colonisation by pioneer bacteria, successive diversification, and changes in microbial population densities until a climax or 'stable' microbiota has established during infancy and early childhood.

The majority of human physiological functions are programmed either in utero, i.e. during pregnancy, or during the early-life window. Thus, the investigators need to determine early-life microbiome profiles over this critical period, particularly what factors influence these microbial signatures, and how changes in the signature are correlated with healthy development during this time-period.

It is proposed that the initial colonisation and establishment of the gut microbiome during early life is closely linked with the promotion of healthy development. Critically, disturbances within this pioneering microbial community (both in mother and baby) have the potential to increase the risk of developing diseases such as autoimmune conditions, allergic-type disorders, infections and chronic intestinal diseases; disturbance may be caused by antibiotics, dietary changes (i.e. breast versus formula milk) and even the way the baby is delivered (i.e. Caesarean section versus vaginal).

The proposed transmission of microbial species from the maternal microbiome to the baby is a key feature of birth, with subsequent waves of colonisation occurring as the baby gets older. There is also an increasing awareness of the importance of maternal health during pregnancy (as affected by obesity and antibiotic use) for the baby's development and health, both before and after birth. Importantly, these life stage events appear to be governed by particular interactions (immune and dietary) that 'select' beneficial microbes such as Bifidobacterium species; species in this genus are prevalent in the gut and vagina of mothers in the later stages of pregnancy and can represent up to 80% of the total microbiome in healthy infants. These pioneering microbe species seem to be important for the development of a healthy microbial community and the subsequent formation of a more 'adult-like' microbiome by the time the child has reached 2-3 years of age; this is thought to be in response to an expanding nutritional environment, i.e. from a milk-based diet to a more complex diet at weaning.

Although several studies have tried to probe these key questions, there are currently many unknowns with respect to this key developmental window including (i) how does the microbiome change in response to different phases of pregnancy across different body sites (and how does this correlate with routinely collected clinical information), (ii) are microbes from mothers directly passed to infants during birth (and how does birth mode affect this i.e. vaginal vs. C-section), (iii) how do factors like diet and antibiotics influence the maternal microbiome, and what is the impact on developing infant microbial communities, (iv) how do different feeding regiments (e.g. breast vs. formula milk) influence specific microbial populations in the infant (e.g. Bifidobacterium), (v) how do these microbes influence immune and metabolic health, and how does this correlate with clinical information captured both in mother and baby over time, and (iv) if the investigators carry out in-depth mechanistic studies using in vitro and in vivo models, can the investigators determine how specific microbes and communities contribute to healthy development and prevent disease incidence?

Critically, if the investigators are to determine the importance of the early life microbiome, the investigators must set-up and carry out comprehensive longitudinal pregnancy and infant studies, i.e. PEARL, to address these key points.

Moreover, gathering these data is critical for implementation of new therapies and health-associated practices that would be expected to have beneficial effects, both in the short-term and across the life course, which could be explored in subsequent studies after PEARL.

The PEARL Study will build on the Chief Investigator's (Hall) ongoing BAMBI Study - Baby Associated Microbiota of the Intestine (University of East Anglia Faculty of Medical Health Research Ethics Committee Reference 2012/2013 - 42 HT), which is collecting faecal samples from preterm infants residing in Neonatal Intensive Care Units (NICUs) and following these babies after they are discharged home for up to 3 years of age. This study has been analysing microbiome signatures in these preterm infants and correlating these to external factors such as antibiotic usage and diet and also immune markers.

ELIGIBILITY:
Inclusion Criteria:

* All participants must be able to understand the requirements of the study and provide signed and dated informed consent for herself and her unborn child.
* Planning to give birth at NNUH or at home.
* At the point of study consent, be ≤22 weeks pregnant.
* BMI between ≥18 - ≤35 kg/m2.
* Must be willing to provide biological samples over a period of 31 months (urine samples, stool samples, low vaginal swabs, skin swabs and breast milk (if breastfeeding this is optional). Blood samples are optional.
* Must be willing to accommodate a small freezer to store frozen samples for the duration of the study.
* Must be willing to complete study questionnaires over a period of 31 months.

Exclusion Criteria:

The participant may not enter the study if ANY of the following apply:

* Pregnancy is for surrogacy purposes.
* Planned adoption, fostering of baby or baby not planned to be living with biological mother.
* Currently taking part in an interventional study.
* Living with or related to a member of the Research Study team.
* Current smoker.
* Taken antibiotics or antifungals or antivirals within the last 3 months. Taken steroids within the last 6 months.
* Currently taking more than a daily dose of probiotics. Have a history of polyps within the gut.
* Have a long-standing gastrointestinal or liver function abnormality requiring on-going medical management or medication.
* Current or history of cancer except for squamous or basal cell carcinomas of the skin that have been medically managed by local excision.
* Unstable dietary history as defined by major changes in diet during the previous month, where participants have stopped or significantly increased a major food group in the diet, for example changed to vegan, vegetarian or stopped eating red meat.
* History of alcohol, drug or substance abuse. Have a history of Hepatitis B or Hepatitis C.
* Any confirmed or suspected pre-existing condition/state of immunosuppression or immunodeficiency (primary or acquired), for example Rheumatoid Arthritis, Type 1 Diabetes, Multiple Sclerosis, Asthma, Eczema and Psoriasis. (Participants who are asymptomatic of Asthma, Eczema and Psoriasis in the last 5 years can be included in the study).
* Major surgery of the gastrointestinal tract, apart from gall bladder or appendix removal, in the past five years.
* Any major bowel resection at any time.
* History of Ulcerative Colitis or Crohn's Disease or Diverticulitis.
* Persistent, infectious gastroenteritis, gastritis, persistent or chronic diarrhoea of unknown cause, Clostridium difficile infection (recurrent) or Helicobacter pylori infection (untreated).
* Chronic constipation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant females less than 22 weeks gestation.
Study Population: 250 pregnant healthy females less than 22 weeks gestation, paired with her newborn baby/babies.
Sampling Method: Non-Probability Sample
Enrollment: 261 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Microbial composition | Baseline and 24 months (11 time points)
  Changes in microbiome measured by DNA/RNA sequencing of longitudinal samples from mothers and their babies.

SECONDARY OUTCOMES:
Microbial signatures identified and correlated with measures of health, host metabolites and immune markers. | Baseline and 24 months (11 time points)
  Changes in microbial composition associated with diet (i.e. breast vs. formula feeding), drugs (i.e.antibiotics), and immune (i.e. cytokine) and metabolites markers measured in paired samples.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Hall, Study Chair — Quadram Institute Bioscience
Locations (1):
- Quadram Institute Bioscience, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Phillips S, Watt R, Atkinson T, Savva GM, Hayhoe A, Hall LJ; PEARL study team. The Pregnancy and EARly Life study (PEARL) - a longitudinal study to understand how gut microbes contribute to maintaining health during pregnancy and early life. BMC Pediatr. 2021 Aug 24;21(1):357. doi: 10.1186/s12887-021-02835-5. PMID 34429088